CLINICAL TRIAL: NCT05591196
Title: Hand and Arm Motor Recovery Via Non-invasive Electrical Spinal Cord Stimulation After Stroke
Acronym: HARNESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chet Moritz, Associate Professor, Electrical and Computer Engineering, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015990
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic; Chronic Stroke
Keywords: Chronic ischemic stroke; Transcutaneous spinal cord stimulation; Activity based rehabilitation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-arm cross-over study: All participants will receive one of the two treatment arms one after the other. The order of the treatments will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Activity Based Rehabilitation (Active Comparator): Activity Based Rehabilitation is comprised of intensive, progressive, functional task practice. The protocol consists of repetitive activities of gross upper limb movement, isolated finger movements, bimanual task performance, simple and complex pinch, and grip performance. Several activities with various difficulty levels are designated for each category, and the participant will perform 1-2 activities within each category in each rehabilitation session. Rehabilitation sessions will be three times per week, 90 minutes per session for six weeks (total of 18 sessions).
  Interventions: Other: Activity Based Rehabilitation
- Non-invasive Electrical Spinal Cord Stimulation + Activity Based Rehabilitation (Experimental): Non-invasive electrical spinal cord stimulation will be performed using surface electrodes placed over the skin of the neck. Biphasic rectangular pulses of 1 millisecond per phase duration will be delivered with a 10 kiloHertz overlapping frequency and between 20-120 Hertzz burst frequency. Non-invasive electrical spinal cord stimulation will be paired with Activity Based Rehabilitation sessions. Stimulation plus rehabilitation sessions will be three times per week, 90 minutes per session for six weeks (total of 18 sessions).
  Interventions: Device: Non-invasive Electrical Spinal Cord Stimulation; Other: Activity Based Rehabilitation

INTERVENTIONS:
Device: Non-invasive Electrical Spinal Cord Stimulation — Electrical stimulation of the spinal cord using surface electrodes
  Arms: Non-invasive Electrical Spinal Cord Stimulation + Activity Based Rehabilitation
Other: Activity Based Rehabilitation — Exercise therapy targeting paralyzed hand and arm

SUMMARY:
The recovery from a stroke is often incomplete. It is the leading cause of acquired permanent disability in the adult population. Persistent functional loss of the hand and arm contributes significantly to disability. However, the current standard of care to treat hand and arm movements are inadequate. There is an urgent need for innovative and effective therapies for recovery of the upper limb after stroke.

Growing evidence shows that electrical spinal cord stimulation, combined with activity-dependent rehabilitation, enables voluntary movement of paralyzed muscles in some neurologic disorders, such as spinal cord injury. The investigators hypothesize that spinal networks that lost control after stroke can be activated by non-invasive electrical stimulation of the spinal cord to improve functional recovery.

The aims of the study are:

1. to determine the improvements in hand and arm function that result from the combined application of non-invasive spinal stimulation and activity-based rehabilitation. Surface electrodes placed over the skin of the neck will be used for non-invasive electrical stimulation of the spinal cord. Functional task practice will be used for activity-dependent rehabilitation,
2. to evaluate long-lasting benefits to hand and arm function that persist beyond the period of spinal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically documented single ischemic stroke resulted in hemiplegia/hemiparesis
* At least six months post-stroke
* Upper Extremity Fugl-Meyer Assessment score "moderate" or "moderate-mild" (29-53 inclusive out of 66) at the screening visit
* Medically and neurologically stable, as determined by medical history and documented physical examination
* For women of childbearing potential, a negative over-the-counter pregnancy test at study entry and willingness to practice adequate contraception during the study
* Ability to attend sessions three times per week
* Adequate social support to participate in all intervention and baseline, follow-up assessment sessions throughout eight months.
* Ability to read, comprehend and speak English

Exclusion Criteria:

* Hemorrhagic stroke
* History of multiple strokes
* Active implanted stimulator (e.g., pacemaker, vagus nerve stimulator, cochlear implant, etc.) or baclofen pump
* Aphasia or any other deficit in communication that interferes with reasonable study participation
* Moderate to severe cognitive impairment
* Presence of neglect (inability to perceive or awareness of, or loss of attention to the weaker half of the body)
* Severe spasticity in the upper limb
* Taking baclofen more than 30 mg/day
* Change in baclofen dose within four weeks before enrollment
* Receiving benzodiazepines, dantrolene, tizanidine, anticoagulant, or antiepileptic medication
* Botulinum toxin injection to the upper limb muscles within six months before enrollment
* Severe joint contractures in the affected hand and arm
* History of spontaneous seizure that had occurred one month or longer after the stroke

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline - Fugl-Meyer assessment of the upper limb | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  The clinician-administered a stroke-specific, performance-based impairment scale. It assesses movement function, sensation, joint range of motion, and pain. The score ranges from 0 to 66. Higher scores indicate better outcomes.
Change from baseline - Pinch and grip force | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  Measurement of hand strengths using a dynamometry.
Change from baseline - Modified Ashworth Scale | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  Clinician-administered test for resistance of a joint to passive movement. This scale grades muscle tone/spasticity. The score ranges from 0 to 4. Higher scores indicate worse outcomes.
Change from baseline - Wolf Motor Function Test | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  Quantifies upper limb motor ability through timed and functional tasks. The score range is 0-75; higher scores denote better function.

SECONDARY OUTCOMES:
Change from baseline - Action Research Arm Test | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  Clinician-administered observational measure to assess upper extremity performance, such as coordination, dexterity, and functioning, in stroke recovery.
Change from baseline - Box and Blocks Test | "Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 8 months."
  Participants move, one by one, the maximum number of blocks from one compartment of a box to another of equal size within 60 seconds. Measures gross manual dexterity.
Change from baseline - Revised Nottingham Sensory Assessment | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  A standardized scale for assessing sensory impairment in stroke patients. Tactile sensation, proprioception, stereognosis, and two-point discrimination are evaluated.
Change from baseline - Stroke Impact Scale | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  A self-report questionnaire that evaluates disability and health-related quality of life after stroke. The questionnaire consists of 8 domains: strength, memory and thinking, emotion, communication, activities of daily living, mobility, hand function, and participation/role function. The score ranges from 0 to 100. Higher scores indicate better outcomes.
Change from baseline - Short Form-36 | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  A self-report health survey questionnaire. The score range from 0 to 100. The higher the score, the better the outcome.
Change from baseline - Patients Global Impression of Change | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  A self-report measure that reflects the participant's belief about the efficacy of treatment: the participant chooses the level of improvement and their functional status between much worse, worse, no change, improved and much improved, compared to the baseline.
Change from baseline - H-reflex test | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  Electrophysiologic evaluation of the reflex response triggered on the motor nerves when sensory fibers in the peripheral nerve are stimulated.
Change from baseline - Somatosensory evoked potentials test | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  Electrophysiologic evaluation of sensory pathways between the brain and the limb.
Change from baseline - Spinally evoked motor potentials test | "Repeated measurements once at baseline, once at the end of each treatment arm and through study completion, an average of 8 months."
  Electrophysiologic evaluation of motor pathways between the central nervous system and the muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Chet Moritz, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No